CLINICAL TRIAL: NCT04853667
Title: Improve Adherence to Weak or Strong Opioid Analgesics at the Time of Care in Children With Hereditary Epidermolysis Bullosa
Acronym: ODEB
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP210420; 2021-A00418-33 (Other: ID RCB number)
Record Dates: First submitted 2021-04-16; First posted 2021-04-21 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Epidermolysis Bullosa
Keywords: Hereditary epidermolysis bullosa (HEB); Pain control; Analgesic treatments
MeSH Terms: conditions — Epidermolysis Bullosa; Agnosia | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients with hereditary epidermolysis bullosa: Minor patients with hereditary epidermolysis bullosa
  Interventions: Other: Interview
- Parents: Parents of patients with hereditary epidermolysis bullosa
  Interventions: Other: Interview

INTERVENTIONS:
Other: Interview — Semi-structured interview, lasting a maximum of one hour

SUMMARY:
Hereditary epidermolysis bullosa (HEB) are rare genodermatoses, clinically characterized by epithelial and subepithelial fragility leading to the formation of blisters and spontaneous erosions on skin at the slightest contact, with possible mucosal damage.

The care of these patients consists of therapeutic baths leading to renew bandages that sometimes covering the entire integument. These are difficult, delicate and painful moments that patients experience daily at home.

For an unexplained reason for 70 to 80% of them, the weak or strong opioid analgesics, deemed necessary and prescribed for good pain control, are not taken on a regular basis as a premedication for baths and dressing changes.

The aim of the study is to understand the child's brakes on taking weak or strong opioid analgesics at the time of care and the parents' difficulties in giving these treatments by means of individual interviews.

DETAILED DESCRIPTION:
Hereditary epidermolysis bullosa (HEB) are rare genodermatoses, clinically characterized by epithelial and subepithelial fragility leading to the formation of blisters and spontaneous erosions on skin at the slightest contact, with possible mucosal damage.

The Pain Medicine and Palliative Medicine Functional Unit (UFMDP) of Necker Hospital is involved on a daily basis in supporting the complex and multidisciplinary management of patients with the most serious forms of hereditary epidermolysis bullosa and their family.

The care of these patients consists of therapeutic baths leading to renew bandages that sometimes covering the entire integument. These are difficult, delicate and painful moments that patients experience daily at home.

The medical and paramedical professionals, from the UFMDP and from the reference center for Genetic Diseases with Cutaneous Expression (MAGEC) (Dermatology Department) of the Necker Hospital, surrounding these children, note that for an unexplained reason for 70 to 80% of them, the weak or strong opioid analgesics, deemed necessary and prescribed for good pain control, are not taken on a regular basis as a premedication for baths and dressing changes.

Care is painful, increasing the vicious circle of anxiety, conflict with caregivers, family and ultimately pain.

The aim of the study is to understand the child's brakes on taking weak or strong opioid analgesics at the time of care and the parents' difficulties in giving these treatments by means of individual interviews.

ELIGIBILITY:
Inclusion Criteria:

* Francophone children and adolescents with hereditary epidermolysis bullosa and of an age to express themselves verbally
* French-speaking holders of parental authority
* Regular follow-ups at the reference center for genetic diseases with cutaneous expression (MAGEC), dermatology department of Necker hospital
* Pain at the time of treatment, the evaluation of which is greater than 4/10 (visual analogue scale VAS) without taking weak or strong opioid analgesics, yet prescribed as premedication
* Holders of parental authority and patients informed and not opposing their participation in the study

Exclusion Criteria:

* Children and adolescents without pain at the time of treatment or for whom paracetamol is sufficient to obtain good pain control
* Children and adolescents already taking analgesic treatments even if their pain is not well balanced at the time of care

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Children and adolescents with hereditary epidermolysis bullosa, follow-ups at the reference center for genetic diseases with cutaneous expression (MAGEC), dermatology department of Necker hospital and their parents.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2021-04-29 (Actual); Primary Completion 2021-05-20 (Actual); Study Completion 2021-05-20 (Actual)

PRIMARY OUTCOMES:
Barriers to taking weak or strong opioid analgesics prescribed | Day 0
  Qualitative analysis of the semi-structured interview

SECONDARY OUTCOMES:
Barriers to giving weak or strong opioid analgesics prescribed | Day 0
  Qualitative analysis of the semi-structured interview

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Chaumon, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Céline Greco, MD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Necker-Enfants Malades, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Understanding noncompliance with opioid-based analgesic premedications in the care of children with hereditary epidermolysis bullosa Authors : Sarah Chaumon, Christine Bodemer, Céline Greco Douleurs : Évaluation - Diagnostic - Traitement Volume 23, Issue 1, February 2022, Pages 14-24